CLINICAL TRIAL: NCT04086472
Title: A Phase 2a Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of MK-1654 in Healthy Participants Inoculated With Experimental Respiratory Syncytial Virus
Brief Title: Phase 2a Respiratory Syncytial Virus (RSV) Human Challenge Study of Clesrovimab (MK-1654) in Healthy Participants (MK-1654-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1654-005; MK-1654-002 (Other: Merck); 2018-003347-28 (EudraCT Number)
Record Dates: First submitted 2019-09-10; First posted 2019-09-11 (Actual); Results first posted 2021-04-13 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Respiratory Syncytial Viruses
MeSH Terms: interventions — MK-1654

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Clesrovimab 100 mg (Experimental): Participants receive a single IV infusion of clesrovimab 100 mg on Day 1.
  Interventions: Biological: Clesrovimab; Biological: RSV-A Memphis 37b
- Clesrovimab 200 mg (Experimental): Participants receive a single IV infusion of clesrovimab 200 mg on Day 1.
  Interventions: Biological: Clesrovimab; Biological: RSV-A Memphis 37b
- Clesrovimab 300 mg (Experimental): Participants receive a single IV infusion of clesrovimab 300 mg on Day 1.
  Interventions: Biological: Clesrovimab; Biological: RSV-A Memphis 37b
- Clesrovimab 900 mg (Experimental): Participants receive a single IV infusion of clesrovimab 900 mg on Day 1.
  Interventions: Biological: Clesrovimab; Biological: RSV-A Memphis 37b
- Placebo (Placebo Comparator): Participants receive a single IV infusion of placebo on Day 1.
  Interventions: Other: Placebo; Biological: RSV-A Memphis 37b

INTERVENTIONS:
Biological: Clesrovimab — Single dose of clesrovimab administered via IV infusion.
  Other Names: MK-1654
  Arms: Clesrovimab 100 mg; Clesrovimab 200 mg; Clesrovimab 300 mg; Clesrovimab 900 mg
Other: Placebo — Placebo (0.9% sodium chloride, USP sterile saline) administered via IV infusion.
  Arms: Placebo
Biological: RSV-A Memphis 37b — Approximately 4Log10 plaque-forming units (PFU)/mL RSV-A virus inoculation strain Memphis 37b administered via intranasal inoculation.

SUMMARY:
The primary objective of this study is to determine if a single intravenous (IV) dose of clesrovimab when administered at 1 of 4 dose levels results in a reduction in viral load after intranasal inoculation (with RSV A Memphis 37b) compared to IV placebo. It is hypothesized that at least 1 of the 4 dose levels of clesrovimab given prior to inoculation will reduce the area under the viral load-time curve (VL-AUC) from Day 2 through Day 11 (inclusive) after viral inoculation (Study Day 31 through Day 40) compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Is a male or female 18 to 55 years of age in good health with no history of major medical conditions that will interfere with participant safety, as defined by medical history, physical examination (including vital signs), electrocardiogram (ECG), and routine laboratory tests and determined by the Investigator at a screening evaluation.
* Has a total body weight ≥ 50 kg and Body Mass Index (BMI) ≥ 18 kg/m^2 and ≤ 30kg/m^2.
* If male, agrees to study contraceptive requirements at dosing and continuing until 90 days after dosing or 28 days after viral inoculation (whichever is later) and to not donate sperm until 90 days after dosing.
* If female, has a negative pregnancy test at screening and prior to dosing and agrees to use one form of highly effective contraception if a woman of childbearing potential (WOCBP), or is not a WOCBP.
* Has serology results within 90 days of dosing that suggest the participant is sensitive to RSV infection (i.e., that they are likely to become infected following inoculation).

Exclusion Criteria:

* Is a female who is breastfeeding or has been pregnant within 6 months prior to enrollment.
* Has a history or evidence of any clinically significant or currently active cardiovascular, respiratory, dermatological, gastrointestinal, endocrinological, haematological, hepatic, immunological (including immune suppression), metabolic, urological, renal, neurological, or psychiatric disease (including participants with a history of depression and/or anxiety with associated severe psychiatric comorbidities.
* Has any significant abnormality altering the anatomy of the nose in a substantial way or nasopharynx that may interfere with the aims of the study and in particular any of the nasal assessments or viral inoculation (historical nasal polyps can be included, but large nasal polyps causing current and significant symptoms and/or requiring regular treatments in the last month will be excluded).
* Has any clinically significant history of epistaxis (large nosebleeds) within the last 3 months prior to IMP dosing and/or history of being hospitalized due to epistaxis on any previous occasion.
* Has a history or currently active symptoms suggestive of upper or lower respiratory tract infection within 6 weeks prior to dosing.
* Has any other major disease that, in the opinion of the Investigator, may interfere with a participant completing the study and necessary investigations.
* Has a history of anaphylaxis-and/or a history of severe allergic reaction or significant intolerance to any food or drug, as assessed by the investigator.
* Has confirmed positive test for drugs of abuse prior to randomization.
* Has a history or presence of alcohol addiction, or excessive use of alcohol (weekly intake in excess of 28 units alcohol; 1 unit being a half glass of beer, a small glass of wine or a measure of spirits), or excessive consumption of xanthine containing substances (e.g. daily intake in excess of 5 cups of caffeinated drinks e.g. coffee, tea, cola).
* Is positive for human immunodeficiency virus (HIV), active hepatitis A (HAV), B (HBV), or C (HCV) test.
* Has evidence of receipt of vaccine within the 4 weeks prior to IMP dosing.
* Has intention to receive any vaccine(s) before the last day of Follow-up.
* Receipt of blood or blood products, or loss (including blood donations) of 470 mL or more of blood during the 3 months prior IMP dosing or planned during the 3 months after the final visit.
* Has use within 7 days prior to IMP dosing of any medication or product (prescription or over-the-counter), for symptoms of hay fever, dermatitis, nasal congestion or respiratory tract infections including the use of regular nasal or dermal corticosteroids or antibiotics, apart from those allowed in the study.
* Has received systemic (intravenous and/or oral) glucocorticoids or systemic antiviral drugs within 6 months prior to IMP dosing.
* Has received chronic (defined as more than 14 continuous days) or current administration of a systemic immunosuppressant or other immune modifying drug, including any dose of oral corticosteroids, within 6 months prior to dose administration. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
* Has used or anticipated use during the conduct of the study of concomitant medications (prescription and/or non-prescription), including vitamins or herbal and dietary supplements within the specified windows (within 7 days prior to IMP dosing), unless in the opinion of the Principal Investigator, the medication will not interfere with the study procedures, outcomes, or compromise participant safety.
* Has a history (participant recall) of receiving any human immunoglobulin preparation
* Has received any investigational drug within 3 months prior to IMP dosing.
* Has received ≥3 investigational drugs within the previous 12 months prior to IMP dosing.
* Has prior participation in another Human Viral Challenge study with a respiratory virus of the same virus family in the preceding 3 months taken from the date of viral challenge in the previous study to the date of expected viral inoculation in this study.
* Has prior participation in any RSV related (vaccine, monoclonal antibody or small molecule) interventional trial.
* Has a forced expiratory volume in 1 second (FEV1) < 80%.
* Has presence of fever, defined as participant presenting with a temperature reading of ≥ 37.9°C on day of IMP dosing.
* Has smoked ≥ 10 pack years at any time [10 pack years is equivalent to one pack of 20 cigarettes a day for 10 years]).
* Has venous access deemed inadequate for the phlebotomy and demands of the study.
* Presents any concern by the investigator regarding safe participation in the study or for any other reason the investigator considers the participant inappropriate for participation in the study.
* Has any contraindication for IV infusion.
* Is or has an immediate family member (eg, spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2020-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- HVIVO Services Ltd ( Site 0001), London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Maas BM, Lommerse J, Plock N, Railkar RA, Cheung SYA, Caro L, Chen J, Liu W, Zhang Y, Huang Q, Gao W, Qin L, Meng J, Witjes H, Schindler E, Guiastrennec B, Bellanti F, Spellman DS, Roadcap B, Kalinova M, Fok-Seang J, Catchpole AP, Espeseth AS, Stoch SA, Lai E, Vora KA, Aliprantis AO, Sachs JR. Forward and reverse translational approaches to predict efficacy of neutralizing respiratory syncytial virus (RSV) antibody prophylaxis. EBioMedicine. 2021 Nov;73:103651. doi: 10.1016/j.ebiom.2021.103651. Epub 2021 Nov 11. PMID 34775220

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult male and female participants were recruited at a single study site in the United Kingdom.
Groups:
- MK-1654 100 mg: Participants receive a single intravenous (IV) infusion of MK-1654 100 mg on Day 1.
- MK-1654 200 mg: Participants receive a single IV infusion of MK-1654 200 mg on Day 1.
- MK-1654 300 mg: Participants receive a single IV infusion of MK-1654 300 mg on Day 1.
- MK-1654 900 mg: Participants receive a single IV infusion of MK-1654 900 mg on Day 1.
Period: Overall Study
Arm/Group | MK-1654 100 mg | MK-1654 200 mg | MK-1654 300 mg | MK-1654 900 mg | Placebo
Started | 16 | 16 | 16 | 16 | 16
Received MK-1654 or Placebo | 16 | 16 | 16 | 16 | 16
Inoculated With Respiratory Syncytial Virus (RSV) A Memphis 37b | 14 | 14 | 14 | 13 | 15
Not Inoculated | 2 | 2 | 2 | 3 | 1
Completed | 12 | 14 | 14 | 13 | 14
Not Completed | 4 | 2 | 2 | 3 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0
Not completed — Various reasons | 2 | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- MK-1654 100 mg: Participants receive a single IV infusion of MK-1654 100 mg on Day 1.
- Total: Total of all reporting groups
Arm/Group | MK-1654 100 mg | MK-1654 200 mg | MK-1654 300 mg | MK-1654 900 mg | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.4 (6.9) | 27.1 (8.3) | 27.6 (8.7) | 26.4 (4.5) | 25.3 (4.1) | 27.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 12 | 5 | 9 | 35
  Male | 12 | 11 | 4 | 11 | 7 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 15 | 16 | 16 | 16 | 16 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1
  White | 14 | 11 | 14 | 15 | 14 | 68
  More than one race | 1 | 2 | 2 | 0 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Viral Load-time Curve (VL-AUC)
Description: The VL-AUC will be determined by reverse transcription qualitative integrated cycler polymerase chain reaction (RT-qPCR) after viral inoculation.
Time Frame: 10 days; from Day 2 through Day 11 (inclusive) after viral inoculation (Study Day 31 through Day 40)
Population: All randomized participants who received a dose of study drug, a RSV inoculation, and had data available are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies-/ml*days
Arm/Group | MK-1654 100 mg | MK-1654 200 mg | MK-1654 300 mg | MK-1654 900 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 14 | 13 | 15
log10 copies-/ml*days | 19.94 [12.11 to 27.78] | 14.74 [6.90 to 22.58] | 16.44 [8.89 to 23.99] | 15.33 [7.50 to 23.17] | 21.25 [13.96 to 28.55]
Statistical Analysis 1: Comparison: MK-1654 100 mg vs Placebo; Treatment vs. Placebo; Test type: Superiority; p = 0.808, ANOVA; Least squares (LS) Mean Difference = -1.31, 90% CI 2-sided [-10.25 to 7.64]
Statistical Analysis 2: Comparison: MK-1654 200 mg vs Placebo; Treatment vs. Placebo; Test type: Superiority; p = 0.229, ANOVA; LS Mean Difference = -6.51, 90% CI 2-sided [-15.46 to 2.43]
Statistical Analysis 3: Comparison: MK-1654 300 mg; Treatment vs. Placebo; Test type: Superiority; p = 0.363, ANOVA; LS Mean Difference = -4.81, 90% CI 2-sided [-13.58 to 3.96]
Statistical Analysis 4: Comparison: MK-1654 900 mg vs Placebo; Treatment vs. Placebo; Test type: Superiority; p = 0.273, ANOVA; LS Mean Difference = -5.92, 90% CI 2-sided [-14.87 to 3.02]

2. Secondary Outcome: Percentage of Participants With Symptomatic Respiratory Syncytial Virus (RSV) Infection
Description: Symptomatic RSV infection is defined as presence of at least 2 quantifiable RT-qPCR at ≥2 consecutive days, plus symptoms of either any grade from 2 different symptoms from the Subject Symptom Card (SSC) or at least one Grade 2 symptom from ≥1 respiratory categories.
Time Frame: 10 days; from Day 2 through Day 11 (inclusive) after viral inoculation (Study Day 31 through Day 40)
Population: All randomized participants who received a dose of study drug, a RSV inoculation, and had data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-1654 100 mg | MK-1654 200 mg | MK-1654 300 mg | MK-1654 900 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 14 | 13 | 15
Percentage of Participants | 53.85 [25.13 to 80.78] | 30.77 [9.09 to 61.43] | 35.71 [12.76 to 64.86] | 30.77 [9.09 to 61.43] | 53.33 [26.59 to 78.73]
Statistical Analysis 1: Comparison: MK-1654 100 mg vs Placebo; Test type: Other — Treatment vs. Placebo; Difference in percentage = 0.51, 95% CI 2-sided [-36.57 to 37.78] — 95% CI based on the Chan and Zhang exact method
Statistical Analysis 2: Comparison: MK-1654 200 mg vs Placebo; Test type: Other — Treatment vs. Placebo; Difference in percentage = -22.56, 95% CI 2-sided [-56.70 to 15.53] — 95% CI based on the Chan and Zhang exact method
Statistical Analysis 3: Comparison: MK-1654 300 mg vs Placebo; Test type: Other — Treatment vs. Placebo; Difference in percentage = -17.62, 95% CI 2-sided [-53.09 to 20.01] — 95% CI based on the Chan and Zhang exact method
Statistical Analysis 4: Comparison: MK-1654 900 mg vs Placebo; Treatment vs. Placebo; Test type: Other — Treatment vs. Placebo; Difference in percentage = -22.56, 95% CI 2-sided [-56.70 to 15.53] — 95% CI based on the Chan and Zhang exact method

3. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 187 days
Population: All participants who received any study intervention are included.
Measure: Number; unit: Participants
Arm/Group | MK-1654 100 mg | MK-1654 200 mg | MK-1654 300 mg | MK-1654 900 mg | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants | 11 | 12 | 12 | 8 | 11

4. Secondary Outcome: Number of Participants With a Serious Adverse Event (SAE)
Description: An SAE is any untoward medical occurrence in a clinical study participant that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event.
Time Frame: Up to 187 days
Population: All participants who received any study intervention are included.
Measure: Number; unit: Participants
Arm/Group | MK-1654 100 mg | MK-1654 200 mg | MK-1654 300 mg | MK-1654 900 mg | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Serum Concentration of MK-1654
Description: The post-dosing concentration of MK-1654 will be determined in serum. On Day 1, 3 samples will be taken at 1, 2, and 4 hours after administration.
Time Frame: Predose and Days 1 (1, 2, and 4 hours postdose), 8, 15, 29, 40, and 57
Population: All randomized participants who received MK-1654 and had no major protocol deviations are included.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | MK-1654 100 mg | MK-1654 200 mg | MK-1654 300 mg | MK-1654 900 mg
Number analyzed (Participants) | 16 | 16 | 16 | 16
µg/mL
  Predose: number analyzed (Participants) | 16 | 15 | 16 | 16
  Predose | 0.0369 (0.148) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 1, 1 hour postdose | 16.4 (3.13) | 36.0 (6.65) | 62.6 (16.8) | 134 (45.1)
  Day 1, 2 hours postdose | 34.3 (6.42) | 72.6 (12.5) | 125 (25.7) | 298 (46.8)
  Day 1, 4 hours postdose | 33.3 (6.19) | 68.8 (11.5) | 122 (26.9) | 287 (46.0)
  Day 8 | 16.0 (2.54) | 33.0 (5.48) | 56.7 (12.8) | 140 (24.1)
  Day 15 | 14.5 (2.49) | 29.1 (4.19) | 47.6 (8.57) | 123 (21.6)
  Day 29: number analyzed (Participants) | 14 | 15 | 14 | 14
  Day 29 | 11.9 (2.11) | 23.1 (3.06) | 38.5 (6.99) | 103 (16.0)
  Day 40: number analyzed (Participants) | 12 | 14 | 14 | 13
  Day 40 | 10.2 (1.74) | 21.4 (3.18) | 35.6 (7.16) | 88.5 (13.4)
  Day 57: number analyzed (Participants) | 11 | 11 | 11 | 8
  Day 57 | 9.46 (2.01) | 18.7 (2.60) | 32.3 (6.14) | 79.5 (15.5)

6. Secondary Outcome: Concentration of RSV Serum Neutralizing Antibody Titers
Description: RSV serum neutralization titers were determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Days 1, 29, 40, and 57
Population: All randomized participants who received a dose of study drug, a RSV inoculation, and had data available for the time point are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MK-1654 100 mg | MK-1654 200 mg | MK-1654 300 mg | MK-1654 900 mg | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Titers
  Day 1, Predose: number analyzed (Participants) | 16 | 15 | 14 | 16 | 15
  Day 1, Predose | 669.1 [487.5 to 918.4] | 699.3 [530.9 to 921.0] | 954.0 [606.1 to 1501.4] | 893.8 [649.0 to 1230.8] | 837.4 [567.9 to 1234.9]
  Day 1, 2 hours postdose: number analyzed (Participants) | 16 | 16 | 15 | 16 | 16
  Day 1, 2 hours postdose | 11137.6 [8884.8 to 13961.7] | 24836.1 [21971.4 to 28074.3] | 41544.8 [33688.4 to 51233.3] | 100163.5 [84649.3 to 118521.1] | 1225.4 [621.0 to 2418.3]
  Day 29: number analyzed (Participants) | 14 | 15 | 14 | 14 | 15
  Day 29 | 4727.2 [4026.3 to 5550.0] | 8135.8 [6945.6 to 9530.0] | 13263.2 [11050.6 to 15918.9] | 31367.8 [26876.0 to 36610.3] | 1037.1 [673.9 to 1596.1]
  Day 40: number analyzed (Participants) | 13 | 14 | 14 | 13 | 15
  Day 40 | 4517.1 [3899.6 to 5232.2] | 8357.6 [7073.1 to 9875.4] | 13510.9 [11564.1 to 15785.4] | 27935.5 [19429.8 to 40164.6] | 1540.4 [1025.9 to 2313.3]
  Day 57: number analyzed (Participants) | 11 | 11 | 11 | 8 | 12
  Day 57 | 4377.8 [3338.4 to 5740.9] | 5531.9 [4315.0 to 7092.1] | 11557.9 [9428.4 to 14168.4] | 22209.6 [17585.6 to 28049.5] | 1500.2 [908.7 to 2476.8]

ADVERSE EVENTS:
Time Frame: Up to 187 days
Description: All participants who received a dose of any study intervention are included.
Arm/Group | MK-1654 100 mg | MK-1654 200 mg | MK-1654 300 mg | MK-1654 900 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 11/16 | 12/16 | 12/16 | 8/16 | 11/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1654 100 mg (N=16) | MK-1654 200 mg (N=16) | MK-1654 300 mg (N=16) | MK-1654 900 mg (N=16) | Placebo (N=16)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (4) | 3 (3) | 1 (1) | 2 (2)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (8) | 6 (6) | 5 (6) | 5 (7) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (7) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT04086472/Prot_SAP_000.pdf